CLINICAL TRIAL: NCT06145711
Title: A Clinical Trial of Parkinson's Disease Treatment by Human-induced Pluripotent Stem Cells (hiPSCs) Derived Dopaminergic Neural Precursor Cells
Brief Title: A Clinical Trial of Parkinson's Disease Treatment by HiPSCs Derived Dopaminergic Neural Precursor Cells
Acronym: hiPSC-DAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XS2022001
Record Dates: First submitted 2023-11-13; First posted 2023-11-24 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease;stem cell
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- to use cell (Experimental)
  Interventions: Other: hiPSC-DAP

INTERVENTIONS:
Other: hiPSC-DAP — Using hiPSC-DAP for the treatment of the patients of Parkinson's diease

SUMMARY:
XellSmart Biomedical (Suzhou) Co., Ltd. has closely collaborated with Shanghai East Hospital(East Hospital Affiliated To Tongji University) , using iPSC seed cells, on the development and establishment of a dopaminergic neural precursor cell production system.

This study is conducted under collaboration between Shanghai East Hospital and XellSmart Biomedical (Suzhou) Co., Ltd. It is a distinctive stem cell therapy research targeting Parkinson's disease patients, characterized by the following:

1. The first instance in China of using autologous iPSC-derived subtype-specific dopaminergic neural precursor cells for alternative transplantation therapy in Parkinson's disease.
2. Before the initiation of this study, there was only one reported case around the world involving the use of laboratory-grade autologous iPSC-induced dopaminergic neural precursor cells for Parkinson's disease treatment in an American Caucasian individual. Positive preliminary clinical research results were obtained and published in the New England Journal of Medicine in 2020. Since then, no similar studies have been reported.

It has great significance to conduct this research. It will fill two critical clinical research gaps in stem cell therapy for Parkinson's disease in the world:

1. The use of clinical-grade autologous iPSCs differentiated into dopaminergic neural cells, and treat Parkinson's disease.
2. Evaluating the safety of using autologous iPSC-differentiated dopaminergic neural cells for Parkinson's disease treatment in individuals of Asian descent or Chinese ethnicity.

DETAILED DESCRIPTION:
This study is a non-randomized, open-label, investigator-initiated interventional clinical trial aimed at exploring the safety of stem cell investigational drugs. The study plans to recruit 3 eligible PD subjects and prepare dopaminergic neural precursor cells from autologous iPSCs in advance. The PD subjects will undergo general anesthesia and, with the assistance of stereotactic technology, receive an injection of autologous iPSC-derived dopaminergic neural precursor cells into the putamen of striatum on one side, transplanted evenly at a linear distance of 1 centimeter. A Sofia drug pouch will also be installed to regularly monitor changes in neurotransmitter metabolism, including dopamine, in the brain.

Following the surgery, there will be regular observations for 6 months, during which the safety of this treatment modality will be examined and analyzed. If the test results within the first 6 months post-surgery indicate both good safety and some level of efficacy, the trial will continue for an additional 6 months. However, if the test results within the first 6 months post-surgery demonstrate good safety (i.e., no adverse events related to stem cell transplantation of grade 3 or higher occurring within 28 days after stereotactic transplantation of dopaminergic neural precursor cells) but insufficient efficacy (evaluated based on subject self-assessment, clinical symptoms, rating scales, PET/MR, changes in the dosage of levodopa, and other medications), autologous iPSC-derived dopaminergic neural precursor cells will be injected into the putamen of striatum on the other side (using the same method). Subsequently, the subjects will be regularly observed for an additional 18 months.

Postoperative observation and follow-up for unilateral stem cell transplantation will be conducted for 12 months, while bilateral stem cell transplantation will be observed and followed for 24 months (with the first postoperative observation and follow-up at 6 months and the second at 18 months). During the study, there will be periodic reviews and summaries every 6 months, generating interim clinical reports to optimize and guide the next stage of data collection and research.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or their legally authorized guardian consents to participate in this study and signs the Informed Consent Form (ICF) in writing.
2. Patients with primary Parkinson's disease, aged between 30 and 70 years, of any gender, with a disease duration of more than 5 years.
3. Hohen-Yahr stage for Parkinson's disease (Appendix V) is between stage 3 and stage 4. Patients with a Hohen-Yahr stage below 3 who refuse other treatments may also be included.
4. The MDS-UPDRS-III score for "OFF" periods in Parkinson's disease is greater than 38 points, and the MDS-UPDRS-III score for the two "OFF" periods before surgery is stable, i.e., (high value - low value) / high value is less than or equal to 10%.
5. Patients who have stably received anti-Parkinson drug therapy for more than 3 months.
6. Previous effective treatment with levodopa, followed by significant drug resistance and wearing-off effect.
7. The patient who is in stable condition, well-controlled complications, no contraindications for general anesthesia, no contraindications for stereotactic surgery, and no other conditions that interfere with clinical assessment.
8. Head MRI does not reveal structural abnormalities that would affect stem cell transplantation, such as severe brain atrophy or space-occupying lesions.
9. Subjects have a caregiver and are able to provide information about their condition before and after stem cell transplantation and can assist the investigator if necessary.

Exclusion Criteria:

1. Patients with atypical Parkinson's disease, such as Parkinson's syndrome or secondary Parkinson's disease.
2. Patients with Parkinson's disease with only tremors.
3. Patients with severe motor impairment preventing the completion of routine motor tasks.
4. Patients with severe neurological deficits caused by other diseases.
5. Patients with severe psychiatric symptoms or dementia.
6. The Patient who is unwilling or unable to cooperate, incapable of self-assessment, and unable to complete assessments even with the help of a physician.
7. Patients who have history of pallidotomy or thalamotomy or deep brain stimulation (DBS) surgery.
8. Patients with apomorphine treatment currently .
9. Coagulation abnormalities (prothrombin time (PT) or international normalized ratio (INR) > 1.5×ULN; activated partial thromboplastin time (APTT) > 1.5×ULN) or receiving anticoagulation therapy.
10. Pregnant or lactating female patients and male and female patients who cannot use effective contraception within 1 year after the last study drug use.
11. Patients who have participated in other drug or medical device clinical studies within the last 3 months.
12. Patients who have used botulinum toxin, phenol, subarachnoid injection of baclofen, or intervention therapy for treating muscle tone disorders or spasticity within the last 6 months.
13. Patients who have history of seizures or prophylactic use of antiepileptic drugs.
14. Patients who have contraindications for general anesthesia or stereotactic surgery, such as sleep apnea or chronic obstructive pulmonary disease, etc.
15. Patients with any other unstable systemic diseases, including active infections, poorly controlled hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg after treatment), unstable angina, congestive heart failure (New York Heart Association NYHA class II or above), or metabolic diseases, etc.
16. Patients with alcohol or drug abuse.
17. Patients who have used a high dose of benzodiazepines within the last 3 months.
18. Patients with severe cognitive impairment, depression, or behavioral disorders, defined as a Mini-Mental State Examination (MMSE) score less than 26 and a Hamilton Depression Rating Scale (HAMD) score greater than 35.
19. History of any malignant tumors.
20. Patients with hepatitis A, active hepatitis B (HBsAg positive with HBV DNA higher than the upper limit of normal, and excluding hepatitis caused by drugs or other reasons), active hepatitis C (anti-HCV antibody positive with HCV RNA higher than the upper limit of normal), hepatitis E, human immunodeficiency virus (HIV) antibody positive, or syphilis (TP antibody positive).
21. Patients with abnormal liver and kidney function laboratory tests during the screening period, such as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3×ULN, serum creatinine >1.5×ULN, or total bilirubin >1.5×ULN.
22. Other situations in which the investigator believes that the subject is not suitable for inclusion or cannot tolerate stem cell transplantation surgery.
23. PD subjects found to have gene mutations by genetic testing.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
1.Number of participants with adverse event (AE), serious adverse event(SAE) and adverse events of special interest(AESI) | 18 Months
  AE occurring throughout the study period will be evaluated using the CTCAE V5.0 standard. AE/SAE and AESI were evaluated after Ommaya sac installation by laboratory examination, measurement of vital signs, physical examination, and subjects' symptoms to detect new abnormalities and/or deterioration of previous conditions and evaluate the safety of the study.
  AESI is defined as intracranial infection, hemorrhage, rejection, and edema within 7 days after Ommaya sac installation, as well as acute allergic reactions and ectopic mass formation associated with study therapy.
  [Time Frame: 18 Months]

SECONDARY OUTCOMES:
Changes in Unified Parkinson's Disease Rating Scale (UPDRS) in OFF state between the experimental group and the control group at 18 months after the first hiPSCs-DAP treatment | day 0, 1 month, 3 month, 6 month, 9 month,12 month,15 month and 18 month
  UPDRS is used for evaluating the impairment and disability associated with Parkinson's Disease (PD). It consists of four sections: (1) Mentation, behavior, and mood; (2) Activities of daily living (ADLs); (3) Motor; and (4) Complications.
  The UPDRS score ranges from 0 to 199, with higher score indicating greater disability [Time Frame: day 0, 1 month, 3 month, 6 month, 9 month,12 month,15 month and 18 month.]
Changes in the Hoehn and Yahr scale | day 0, 1 month, 3 month, 6 month, 9 month,12 month,15 month and 18 month
  Hoehn and Yahr scale is used to provide a general estimate of clinical function of PD patients, combining functional deficits (disability) and objective signs (impairment). The Hoehn and Yahr score ranges from 0 to 5, with higher score indicating higher dysfunction of PD patients
Changes in the Schwab and England score | day 0, 1 month, 3 month, 6 month, 9 month,12 month,15 month and 18 month
  The Schwab and England score develop a scale that describes the capacity of daily living shown by a PD patients. It measures the following three areas: dependence, abilities, and awareness. The Schwab and England score range from o% to 100%, with higher scores indicating greater healthy status.
Changes in the Parkinson's Disease Questionnaire (PDQ-39) | day 0, 1 month, 3 month, 6 month, 9 month,12 month,15 month and 18 month
  PDQ-39 provides the evidence of the quality of life of a PD patient. The higher the score, the lower the quality of life of PD patients.
Hamilton Depression Rating Scale (HAM-D) | day 0, 1 month, 3 month, 6 month, 9 month,12 month,15 month and 18 month
  HAMD is the most widely used scale in clinical evaluation of depression in PD patients. This project takes 8 points as the critical value of depression, and the total score over 35 points is considered as severe depression, more than 20 points is likely to be diagnosed with depression, less than 8 points is not depressed.
Cranial dopamin transporter measured by positron emission tomography (PET)- magnetic resonance imaging (MRI) | [Time Frame: 3 month, 6 month, 18 month]
  Changes of cranial expression of dopamine transporter investigated by PET-M

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided